CLINICAL TRIAL: NCT05082116
Title: A Multi-centre, Open-label Trial Evaluating Efficacy, Safety and Pharmacokinetics of Turoctocog Alfa Pegol (N8-GP) When Used for Treatment and Prophylaxis of Bleeding Episodes in Previously Treated Chinese Patients With Haemophilia A
Brief Title: Efficacy and Safety of Turoctocog Alfa Pegol (N8-GP) for Prophylaxis and Treatment of Bleeding Episodes in Previously Treated Chinese Patients With Haemophilia A (pathfinder10)
Acronym: Pathfinder10
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NN7088-4595; U1111-1235-5905 (Other: World Health Organization (WHO)); 2020-003001-58 (EudraCT Number)
Record Dates: First submitted 2021-09-21; First posted 2021-10-18 (Actual); Results first posted 2024-01-18 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Haemophilia A
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- N8-GP prophylaxis (Experimental): All patients will receive prophylaxis with 50 IU/kg N8-GP every 4 days for a treatment period of at least 28 weeks (with the possibility of switching to twice-weekly dosing during the treatment period at the discretion of the investigator).
  Interventions: Drug: turoctocog alfa pegol (N8-GP)

INTERVENTIONS:
Drug: turoctocog alfa pegol (N8-GP) — N8-GP will be injected into a vein (intravenous injections) every 4 days in at least 28 weeks

SUMMARY:
The study investigates how well the medicine called turoctocog alfa pegol (N8-GP) works in previously treated Chinese patients with severe haemophilia A.

Participants will be treated with N8-GP. This is a medicine that doctors can already prescribe in other countries.

The medicine will be injected into a vein (intravenous injections) and blood samples will be collected.

The study will last for about 7-8 months. Participants will have between 8 and 15 visits to the clinic and possibly a number of phone calls with the study doctor.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any trial-related activities. Trial-related activities are any procedures that are carried out as part of the trial, including activities to determine suitability for the trial.
* Male Chinese patient with severe congenital haemophilia A with a FVIII activity below 1% according to medical records.
* Aged greater than or equal to 12 years at the time of signing informed consent.
* History of at least 150 exposure days (EDs) to other FVIII products.
* The patient and/or caregiver is capable of assessing a bleeding episode, keeping a diary, performing home treatment of bleeding episodes and otherwise following the trial procedures at the discretion of the investigator.

Exclusion Criteria:

* Known or suspected hypersensitivity to trial product or related products.
* Previous participation in this trial. Participation is defined as signed informed consent.
* Participation in any clinical trial of an approved or non-approved investigational medicinal product within 5 half-lives or 30 days from screening, whichever is longer.
* Known history of FVIII inhibitors based on existing medical records, laboratory report reviews and patient and/or caregiver interviews.
* Current FVIII inhibitors greater than or equal to 0.6 BU.
* Congenital or acquired coagulation disorder other than haemophilia According to medical records.
* HIV positive, defined by medical records, with CD4+ count less than or equal 200/L and a viral load greater than 200 particles/μl or greater than 400000 copies/mL within 6 months of the trial entry. If the data are not available in medical records within last 6 months, then the test must be performed at screening visit.
* Previous significant thromboembolic events (e.g. myocardial infarction, cerebrovascular disease or deep venous thrombosis) as defined by available medical records.
* Hepatic dysfunction defined as aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) greater than 3 times limit of normal combined with total bilirubin greater than 1.5 times the upper limit of normal at screening, as defined by central laboratory
* Renal impairment defined as estimated glomerular filtration rate (eGFR) below or equal to 30 mL/min/1.73 m^2 for serum creatinine measured at screening, as defined by central laboratory.
* Platelet count below 50×109/L at screening based on central laboratory values at screening.
* Ongoing immune modulating or chemotherapeutic medication.
* Any disorder, except for conditions associated with haemophilia A, which in the investigator's opinion might jeopardise the patient's safety or compliance with the protocol.
* Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation.

Min Age: 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2021-09-27 (Actual); Primary Completion 2022-12-28 (Actual); Study Completion 2022-12-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 1452), Study Director — Novo Nordisk A/S
Locations (11):
- China (11):
  - Beijing Children's Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Fujian Medical University Union Hospital-Hematology, Fuzhou, Fujian
  - Nanfang Hospital, Southern Medical University-Haematology, Guangzhou, Guangdong
  - The Affiliated Hospital of Guizhou Medical University-Hematology, Guiyang, Guizhou
  - Xiangya Hospital Central-South University, Changsha, Hunan
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Qinghai Provincial People's Hospital, Xining, Qinghai
  - Jinan Central Hospital, Jinan, Shandong
  - Institute of Hematology and Blood Diseases Hospital, Tianjin-Hematology, Tianjin, Tianjin Municipality
  - Institute of hematology and Blood Diseases Hospital, Tianjin, Tianjin, Tianjin Municipality
  - The Second Affiliated Hospital of Kunming Medical University, Kunming, Yunnan

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 36 Chinese participants with a severe haemophilia A were recruited in this trial. The trial was conducted at 8 sites in China mainland.
Groups:
- Adolescents (12-17 Years): Participants with haemophilia A aged 12-17 years with greater than or equal to (≥) 150 exposure days to other FVIII product received one single bolus dose of 50 international unit per Kilogram (IU/kg) of turoctocog alfa pegol (N8-GP), administered intravenously (IV) every 4th day (96 hours) or twice weekly (investigator's discretion). All bleeds were to be treated with doses between 20-75 IU/kg according to the severity and location of the bleeding episode.
- Adults (18-70 Years): Participants with haemophilia A aged 18-70 years with ≥150 exposure days to other FVIII product received one single bolus dose of 50 IU/kg of turoctocog alfa pegol (N8-GP), administered IV every 4th day (96 hours) or twice weekly (investigator's discretion). All bleeds were to be treated with doses between 20-75 IU/kg according to the severity and location of the bleeding episode.
Period: Overall Study
Arm/Group | Adolescents (12-17 Years) | Adults (18-70 Years)
Started | 13 | 23
Full Analysis Set | 13 | 23
Safety Analysis Set | 13 | 23
Pharmacokinetic (PK) Analysis Set | 4 | 11
Completed | 13 | 23
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Results were based on the full analysis set (FAS) which included all participants exposed to N8-GP in this trial.
Groups:
- Total: Total of all reporting groups
Arm/Group | Adolescents (12-17 Years) | Adults (18-70 Years) | Total
Number analyzed (Participants) | 13 | 23 | 36
Age, Continuous [Mean (Standard Deviation); unit: Years] | 13.7 (1.7) | 28.7 (9.2) | 23.3 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 13 | 23 | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 13 | 23 | 36
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 13 | 23 | 36
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Bleeding Episodes Per Year (Annualised Bleeding Rate)
Description: Number of bleeding episodes per year (Annualised Bleeding Rate) data is reported. Annualised bleeding rate (ABR) is the number of bleeding episodes per year.
Time Frame: From start of treatment (Week 0) until Week 28
Population: Results were based on the FAS which included all participants exposed to N8-GP in this trial.
Measure: Median (Inter-Quartile Range); unit: Bleeding episodes per year
Arm/Group | Adolescents (12-17 Years) | Adults (18-70 Years)
Number analyzed (Participants) | 13 | 23
Bleeding episodes per year | 0.00 [0.00 to 1.63] | 0.00 [0.00 to 1.83]

2. Secondary Outcome: Haemostatic Effect of N8-GP When Used for Treatment of Bleeding Episodes, Assessed on a Four-point Scale for Haemostatic Response (Excellent, Good, Moderate and None)
Description: Haemostatic effect of N8-GP for treatment of bleeding episodes was assessed by 4-point response scale: none, moderate, good or excellent. Evaluation during trial was done by participant and/or parent(s)/caregiver within approximately 8 hours after a single injection as follows: Excellent: Abrupt pain relief and/or clear improvement in objective signs of bleeding within approximately 8 hrs after a single injection; Good: Definite pain relief and/or improvement in signs of bleeding within approximately 8 hrs after a single injection, but possibly requiring more than one injection for complete resolution; Moderate: Probable or slight beneficial effect within approximately 8 hours after the first injection, but usually requiring more than one injection; None: No improvement, or worsening of symptoms.
Time Frame: From start of treatment (Week 0) until Week 28
Population: Results were based on the FAS which included all participants exposed to N8-GP in this trial.
Measure: Number; unit: Bleeding Episodes
Arm/Group | Adolescents (12-17 Years) | Adults (18-70 Years)
Number analyzed (Participants) | 13 | 23
Bleeding Episodes
  Excellent | 18 | 22
  Good | 3 | 6
  Moderate | 3 | 0
  None | 0 | 0
  Missing | 0 | 0

3. Secondary Outcome: Number of Injections Needed to Treat Bleeding Episodes
Description: The mean number of injections of N8-GP used for treatment of a bleed from start to stop of a bleed was reported.
Time Frame: From start of treatment (Week 0) until Week 28
Population: Results were based on the FAS which included all participants exposed to N8-GP in this trial.
Measure: Mean (Standard Deviation); unit: Injections per bleed
Units Other Than Participants: Bleeding episodes
Arm/Group | Adolescents (12-17 Years) | Adults (18-70 Years)
Number analyzed (Participants) | 13 | 23
Number analyzed (Bleeding episodes) | 24 | 28
Injections per bleed | 2 (0.8) | 1 (0.3)

4. Secondary Outcome: Consumption of N8-GP for Prophylaxis
Description: The mean consumption of N8-GP for prophylaxis per year per participant was reported and it was measured in international units per kilogram per year (IU/kg/year).
Time Frame: From start of treatment (Week 0) until Week 28
Population: Results were based on the FAS which included all participants exposed to N8-GP in this trial.
Measure: Mean (Standard Deviation); unit: IU/kg/year
Arm/Group | Adolescents (12-17 Years) | Adults (18-70 Years)
Number analyzed (Participants) | 13 | 23
IU/kg/year | 4909.5 (252.0) | 4873.9 (237.6)

5. Secondary Outcome: FVIII Trough Activity During Prophylaxis
Description: Trough levels of FVIII was reported for all participnats who received prophylaxis treatment. Chromogenic assay was performed with N8-GP product specific standard (PSS) as a calibrator. The analysis is based on a mixed model on the log transformed plasma FVIII activity with age group as fixed effect and participant as a random effect. The mean trough is presented back-transformed to the natural scale.
Time Frame: From start of treatment (Week 0) (excluding the first exposure) until Week 28
Population: Results were based on the FAS which included all participants exposed to N8-GP in this trial.
Measure: Mean (95% Confidence Interval); unit: International unit per milliliter(IU/mL)
Arm/Group | Adolescents (12-17 Years) | Adults (18-70 Years)
Number analyzed (Participants) | 13 | 23
International unit per milliliter(IU/mL) | 0.032 [0.023 to 0.044] | 0.034 [0.025 to 0.045]

6. Secondary Outcome: Percentage of Participants With Incidence Rate of Confirmed FVIII Inhibitors ≥0.6 BU
Description: Percentage of participants who developed inhibitory antibodies against FVIII was presented. A participant was said to have FVIII-inhibitors if two consecutive tests, preferably within 2 weeks, were positive (greater than or equal to (≥) 0.6 bethesda unit (BU)). For the calculation of the inhibitor rate the numerator was included for all participants with neutralising antibodies while the denominator was included for all participants with a minimum of 50 exposures plus any participants with less than 50 exposures but with neutralising inhibitor.
Time Frame: From start of treatment (Week 0) until Week 28
Population: Results were based on the FAS which included all participants exposed to N8-GP in this trial.
Measure: Number; unit: Percentage of participants
Arm/Group | Adolescents (12-17 Years) | Adults (18-70 Years)
Number analyzed (Participants) | 13 | 23
Percentage of participants | 0.00 | 0.00

7. Secondary Outcome: Number of Adverse Events (AEs)
Description: An adverse event (AE) was defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom or disease temporally associated with the use of a product, whether or not considered related to the product. All presented AEs are treatment-emergent. A treatment-emergent adverse event was defined as an event with onset after first N8-GP administration.
Time Frame: From start of treatment (Week 0) until end of trial (Week 32)
Population: Results were based on the safety analysis set (SAS) which included all participants exposed to N8-GP in this trial.
Measure: Number; unit: Events
Arm/Group | Adolescents (12-17 Years) | Adults (18-70 Years)
Number analyzed (Participants) | 13 | 23
Events | 15 | 25

8. Secondary Outcome: Number of Serious Adverse Events (SAEs)
Description: A serious adverse event (SAE) is defined as any untoward medical occurrence that at any dose results in death, or is life-threatening, or requires inpatient hospitalization or causes prolongation of existing hospitalization results in persistent or significant disability/incapacity, or may have caused a congenital anomaly/birth defect, or requires intervention to prevent permanent impairment or damage. All presented SAEs are treatment-emergent (any serious adverse events which occurred after trial product administration).
Time Frame: From start of treatment (Week 0) until end of trial (Week 32)
Population: Results were based on the SAS which included all participants exposed to N8-GP in this trial.
Measure: Number; unit: Events
Arm/Group | Adolescents (12-17 Years) | Adults (18-70 Years)
Number analyzed (Participants) | 13 | 23
Events | 0 | 0

9. Secondary Outcome: Incremental Recovery (IR)
Description: The incremental recovery was calculated by subtracting the FVIII activity (IU/mL) measured in plasma at time 0 from that measured at time 30 min after dosing and dividing this difference by the dose injected at time 0 expressed as IU/kg body weight. FVIII activity was measured with a chromogenic assay.
Time Frame: 30 min post-injection at Week 0, Week 28
Population: The PK analysis set included sub-set of participants from FAS who were included for PK assessments. Number analyzed = Number of participants with available data for specific timepoints.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (IU/mL)/(IU/kg)
Arm/Group | Adolescents (12-17 Years) | Adults (18-70 Years)
Number analyzed (Participants) | 4 | 11
(IU/mL)/(IU/kg)
  Week 0: number analyzed (Participants) | 4 | 10
  Week 0 | 0.023 (28.107) | 0.023 (28.367)
  Week 28: number analyzed (Participants) | 3 | 11
  Week 28 | 0.029 (1.443) | 0.024 (23.535)

10. Secondary Outcome: FVIII Activity 30 Min Post-injection (C30min)
Description: FVIII plasma activity was measured after 30 mins of injection. FVIII activity was measured with a chromogenic assay.
Time Frame: 30 min post-injection at Week 0, Week 28
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: IU/mL
Arm/Group | Adolescents (12-17 Years) | Adults (18-70 Years)
Number analyzed (Participants) | 4 | 11
IU/mL
  Week 0: number analyzed (Participants) | 4 | 10
  Week 0 | 1.178 (24.531) | 1.196 (27.304)
  Week 28: number analyzed (Participants) | 3 | 11
  Week 28 | 1.557 (0.646) | 1.302 (21.521)

11. Secondary Outcome: FVIII Trough Activity 96 h Post-injection (C96h)
Description: FVIII plasma activity was measured after 96 h of injection. This was measured at two time points Week 0 and Week 28 during the study. Chromogenic assay was performed.
Time Frame: Single-dose: 96 h ± 8 h post-injection at Week 0, Steady-state: 96 h ± 8 h post-injection at Week 28
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: IU/mL
Arm/Group | Adolescents (12-17 Years) | Adults (18-70 Years)
Number analyzed (Participants) | 4 | 11
IU/mL
  Week 0: number analyzed (Participants) | 4 | 10
  Week 0 | 0.033 (36.048) | 0.039 (44.608)
  Week 28: number analyzed (Participants) | 3 | 11
  Week 28 | 0.032 (14.616) | 0.045 (58.020)

12. Secondary Outcome: Area Under the Curve (AUC0-inf)
Description: Area under the plasma activity versus time profile from time zero to infinity (AUC0-inf) was measured.
Time Frame: 0-96 hours post-injection at Week 0 and Week 28
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*(IU/mL)
Arm/Group | Adolescents (12-17 Years) | Adults (18-70 Years)
Number analyzed (Participants) | 4 | 11
h*(IU/mL)
  Week 0: number analyzed (Participants) | 4 | 10
  Week 0 | 31.556 (20.100) | 33.650 (26.123)
  Week 28: number analyzed (Participants) | 3 | 11
  Week 28 | 37.274 (4.541) | 37.952 (28.030)

13. Secondary Outcome: Area Under the Curve (0-t)
Description: Area under the plasma activity versus time profile from time zero to last measurable activity (AUC0-t) was measured.
Time Frame: 0-96 hours post-injection at Week 0 and Week 28
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*(IU/mL)
Arm/Group | Adolescents (12-17 Years) | Adults (18-70 Years)
Number analyzed (Participants) | 4 | 11
h*(IU/mL)
  Week 0: number analyzed (Participants) | 4 | 10
  Week 0 | 30.578 (19.999) | 32.300 (26.565)
  Week 28: number analyzed (Participants) | 3 | 11
  Week 28 | 36.467 (4.292) | 36.406 (27.173)

14. Secondary Outcome: Area Under the Curve (0-96h)
Description: Area under the plasma activity versus time profile from time zero to 96 hours (AUC0-96h) was measured.
Time Frame: 0-96 hours post-injection at Week 0 and Week 28
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*(IU/mL)
Arm/Group | Adolescents (12-17 Years) | Adults (18-70 Years)
Number analyzed (Participants) | 4 | 11
h*(IU/mL)
  Week 0: number analyzed (Participants) | 4 | 10
  Week 0 | 30.509 (19.989) | 32.269 (26.558)
  Week 28: number analyzed (Participants) | 3 | 11
  Week 28 | 36.428 (4.251) | 36.398 (27.168)

15. Secondary Outcome: Accumulation Ratio
Description: Accumulation ratio was calculated as AUC(0-96h) at steady state/AUC(0-96h) at single dose. AUC(0-96) is the area under the plasma activity versus time profile from time zero to 96 hours.
Time Frame: 0-96 hours post-injection on Week 28
Population: The PK analysis set included sub-set of participants from FAS who were included for PK assessments. Overall number of partianalyzed = Number of participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of AUC
Arm/Group | Adolescents (12-17 Years) | Adults (18-70 Years)
Number analyzed (Participants) | 3 | 10
Ratio of AUC | 1.152 (19.682) | 1.086 (53.085)

16. Secondary Outcome: Terminal Half-life (t½)
Description: Terminal half life was calculated as ln(2)/λz; where λz is the terminal elimination rate constant. The terminal elimination rate constant was estimated using linear regression on the terminal part of the log (activity) versus time profile.
Time Frame: 0-96 hours post-injection on Week 0 and Week 28
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour (h)
Arm/Group | Adolescents (12-17 Years) | Adults (18-70 Years)
Number analyzed (Participants) | 4 | 11
hour (h)
  Week 0: number analyzed (Participants) | 4 | 10
  Week 0 | 19.106 (14.019) | 20.200 (20.422)
  Week 28: number analyzed (Participants) | 3 | 11
  Week 28 | 17.729 (5.568) | 20.238 (18.882)

17. Secondary Outcome: Clearance (CL)
Description: Clearance (CL) of drug after intravenous administration was reported. Clearance was calculated using the formula CL= Dose / AUC(0-inf) for single dose and CL= Dose / AUC(0-96) h for steady state.
Time Frame: Single-dose: 0-96 h post-injection at Week 0, Steady-state: 0-96 h post-injection at Week 28
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milliter per hour per kilogram (mL/h/kg)
Arm/Group | Adolescents (12-17 Years) | Adults (18-70 Years)
Number analyzed (Participants) | 4 | 11
milliter per hour per kilogram (mL/h/kg)
  Week 0: number analyzed (Participants) | 4 | 10
  Week 0 | 1.636 (17.092) | 1.550 (29.123)
  Week 28: number analyzed (Participants) | 3 | 11
  Week 28 | 1.434 (4.488) | 1.434 (25.335)

18. Secondary Outcome: Apparent Volume of Distribution (Vz) Based on the Terminal Phase
Description: Apparent volume of distribution (Vz) based on the terminal phase was measured. Apparent volume of distribution was calculated using formula: total plasma clearance divided by terminal elimination rate constant (Vz= CL/λz).
Time Frame: 0-96 hours post-injection on Week 0 and Week 28
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milliter per kilogram (mL/kg)
Arm/Group | Adolescents (12-17 Years) | Adults (18-70 Years)
Number analyzed (Participants) | 4 | 11
milliter per kilogram (mL/kg)
  Week 0: number analyzed (Participants) | 4 | 10
  Week 0 | 45.098 (24.375) | 45.165 (34.649)
  Week 28: number analyzed (Participants) | 3 | 11
  Week 28 | 36.673 (4.042) | 41.878 (27.534)

19. Secondary Outcome: Apparent Volume of Distribution (Vss) Based on Steady-state
Description: Apparent volume of distribution (Vss) at steady-state was measured. Apparent volume of distribution (Vss) was calculated using formula: total plasma clearance multiplied by mean residence time (Vss=CL*MRT).
Time Frame: 0-96 h post-injection at Week 28
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milliter per kilogram (mL/kg)
Arm/Group | Adolescents (12-17 Years) | Adults (18-70 Years)
Number analyzed (Participants) | 3 | 11
milliter per kilogram (mL/kg) | 34.511 (5.727) | 39.786 (28.558)

20. Secondary Outcome: Extrapolated Area Under the Curve (AUC Percent [%] Extrap
Description: Percentage of AUC(0-inf) determined by extrapolation. It was calulating using formula: Area under the plasma activity versus time profile from given measurable time to infinity (AUCt-inf)/Area under the plasma activity versus time profile from time zero to infinity (AUC0-inf).
Time Frame: 0-96 hours post-injection on Week 0 and Week 28
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of AUC
Arm/Group | Adolescents (12-17 Years) | Adults (18-70 Years)
Number analyzed (Participants) | 4 | 11
Percentage of AUC
  Week 0: number analyzed (Participants) | 4 | 10
  Week 0 | 2.847 (47.917) | 3.392 (63.420)
  Week 28: number analyzed (Participants) | 3 | 11
  Week 28 | 2.143 (17.743) | 3.424 (65.849)

21. Secondary Outcome: Mean Residence Time
Description: Mean residence time (MRT) calculated as area under the first moment plasma concentration-time curve (AUMC [0-inf]) divided by AUC (0-inf). (AUMC [0-inf]) is the area under the first moment plasma concentration-time curve from time 0 to infinity.
Time Frame: 0-96 hours post-injection on Week 0 and Week 28
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour
Arm/Group | Adolescents (12-17 Years) | Adults (18-70 Years)
Number analyzed (Participants) | 4 | 11
hour
  Week 0: number analyzed (Participants) | 4 | 10
  Week 0 | 27.101 (13.400) | 27.941 (21.114)
  Week 28: number analyzed (Participants) | 3 | 11
  Week 28 | 24.070 (4.347) | 27.739 (22.177)

22. Secondary Outcome: Terminal Elimination Rate Constant (λz)
Description: The terminal elimination rate constant was estimated using linear regression on the terminal part of the log(activity) versus time profile.
Time Frame: 0-96 hours post-injection on Week 0 and Week 28
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/hour
Arm/Group | Adolescents (12-17 Years) | Adults (18-70 Years)
Number analyzed (Participants) | 4 | 11
1/hour
  Week 0: number analyzed (Participants) | 4 | 10
  Week 0 | 0.036 (13.526) | 0.034 (18.083)
  Week 28: number analyzed (Participants) | 3 | 11
  Week 28 | 0.039 (5.749) | 0.034 (16.862)

ADVERSE EVENTS:
Time Frame: From start of treatment (Week 0) until end of trial (Week 32)
Description: All presented AEs are treatment-emergent adverse events. A TEAEs was defined as an event with onset after first N8-GP administration. Results were based on the SAS which included all participants exposed to N8-GP in this trial.
Arm/Group | Adolescents (12-17 Years) | Adults (18-70 Years)
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/23
Other Adverse Events (participants affected / at risk) | 7/13 | 4/23
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adolescents (12-17 Years) (N=13) | Adults (18-70 Years) (N=23)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Medication error (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (2) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.

DOCUMENTS (2):
  • Study Protocol (2021-07-05): https://cdn.clinicaltrials.gov/large-docs/16/NCT05082116/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-29): https://cdn.clinicaltrials.gov/large-docs/16/NCT05082116/SAP_001.pdf